CLINICAL TRIAL: NCT01726959
Title: Prediction of Methotrexate Response - A Pilot Study
Acronym: MRS
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: MRS1
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2015-08

CONDITIONS: Rheumatoid Arthritis; Rheumatic Diseases
Keywords: methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Methotrexate: Methotrexate for rheumatic diseases, 2.5 - 25 mg weekly

SUMMARY:
The objective of this study is to identify genetic predictors of individual methotrexate (MTX) response in patients with rheumatic diseases by determining genetic and metabolomic factors related to nutrient metabolism and drug transport.

The development of better genetic predictors of individual MTX treatment response would provide invaluable prognostic information prior to initiating treatment, which would allow more appropriate choice of therapy, decreased adverse events, and more efficient dose-escalation of the drug, with ultimate benefits of improved effectiveness and tolerability rates in patients being treated with MTX for autoimmune diseases.

Despite being the gold-standard therapy for rheumatoid arthritis and other types of chronic autoimmune diseases since 1951, MTX's efficacy and safety profile limit its use: MTX is discontinued in greater than 50% of patients secondary to inefficacy or poor tolerability. Upon initial treatment, discontinuation rates approach 12% because of drug toxicity, despite prophylactic measures such as the co-administration of folic acid. The causes of primary failure, secondary failure, and adverse events of MTX may be related to genetic variation of dihydrofolate reductase (DHFR) and other genes involved in folate metabolism, one-carbon transfer, and drug transport. The purpose of this study is to identify genetic variations involved in methotrexate response so that we may better understand the pharmacodynamics of MTX metabolism in patients with rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (i.e. >18 years of age) who are enrolled at NorthEast Rheumatology at the Carolinas Medical Center - NorthEast who will be initiating MTX as standard treatment for their particular rheumatic disease, which may include (but not be limited to) conditions such as rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, inflammatory-bowel disease related arthropathies, lupus (systemic lupus erythematosus, cutaneous lupus erythematosus), Sjogren's syndrome, Behcet's disease, systemic sclerosis, and vasculitides.
* No prior enrollment into this study
* Enrollment and initial blood sample collection prior to first MTX administration
* Written informed consent

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with rheumatic disease being newly treated with methotrexate, recruited from a single rheumatology practice
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
lymphocyte proliferation | 9 days in culture

SECONDARY OUTCOMES:
dihydrofolate reductase expression | 9 days in culture

CONTACTS AND LOCATIONS:
Overall Officials: Gordon K. Lam, MD, Principal Investigator — Carolinas Medical Center - NorthEast Rheumatology
Locations (1):
- Carolinas Medical Center - NorthEast, Concord, North Carolina, United States